CLINICAL TRIAL: NCT02072707
Title: Prospective and Randomized Study to Evaluate Efficacy and Safety of Epicardial Ventricular Tachycardia Ablation Using Contact Force Sensor Irrigated Tip Catheter - Pilot Study
Brief Title: Efficacy and Safety of Epicardial VT Ablation Using Contact Force Irrigated Tip Catheter - Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Arrhythmia Clinical Unit Director, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Arrit-Incor-1
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Tachycardia, Ventricular
Keywords: Ventricular Tachycardia; RF ablation; Epicardial Access; Contact Sensor Irrigated tip catheter
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epicardial VT ablation (Active Comparator): Patients will underwent combined epicardial and endocardial mapping and ablation
  Interventions: Procedure: Epicardial VT ablation
- Endocardial VT Ablation (Active Comparator): Patients will underwent endocardial only VT mapping and ablation
  Interventions: Procedure: Endocardial VT Ablation

INTERVENTIONS:
Procedure: Epicardial VT ablation — Combined Epicardial and Endocardial VT Ablation
  Arms: Epicardial VT ablation
Procedure: Endocardial VT Ablation — Endocardial Only VT ablation
  Arms: Endocardial VT Ablation

SUMMARY:
The investigators hypothesized that combined endocardial and epicardial VT ablation using contact sensor irrigated catheter is safe and achieves a lower recurrence rate than endocardial only ablation in ischemic and non-ischemic patients, for this the investigators will randomize 20 patients in two groups, one with endocardial only ablation and other with combined endocardial and epicardial ablation.

DETAILED DESCRIPTION:
Pilot Study Design The investigators will select 20 ischemic or non-ischemic cardiomyopathy patients with scar related Ventricular tachycardia with indication of VT ablation. After informed consent, these patients will be randomized to endocardial only (Control Group) or combined endocardial and epicardial ablation (Treatment Group).

Inclusion Criteria Patients with ischemic and non-ischemic cardiomyopathy and recurrent sustained monomorphic VT requiring cardioversion or antiarrhythmic drug administration with ≥4 episodes in the previous 6 months despite an ICD or antiarrhythmic drug therapy. Patients without ICD were eligible after 2 episodes of sustained VT.

Exclusion Criteria Creatinine level >2.5mg/dL; LV ejection fraction <10%; NYHA Class IV; mobile thrombus on LV; absence of vascular access to the LV; life-expectancy of less than 12 months; previous open-chest cardiac surgical procedure; unstable angina; myocardial infarction in the last 2 months; severe aortic stenosis; severe mitral regurgitation secondary to leaflet or chordae rupture; pregnancy and age of less than 18 years old.

Ablation Technique In the patients randomized for combined epicardial and endocardial ablation, subxyphoid puncture will be performed according to previously described technique. Following successful epicardial access on the combined epi and endocardial ablation and following the venous puncture on the endocardial only group, a puncture of femoral artery will be performed. If the patient has peripheral artery disease, the catheter will be positioned on the left ventricle through transeptal puncture.

Electroanatomic voltage map will be constructed of the endocardial and epicardial surface. After map construction, programmed ventricular stimulation of the apex of the RV with S4 extrastimuli will be performed aiming for VT inducibility. If the induced VT is well tolerated, activation mapping of the VT will be constructed in addition to entrainment mapping. If the VT is not hemodynamically tolerated, it will be reverted either by Burst or electrical cardioversion, than substrate modification in the scar combined with pace-mapping and local abnormal electrograms (late potentials) ablation will be performed. In the patients in the endocardial only group, only the endocardial surface of the right or left ventricle will be ablated.

In the combined epicardial and endocardial group, the choice of the surface to be ablated will be guided by the tachycardia mapping (mesodiastolic and pre-systolic potentials), extension of the scar, pace-mapping in both surfaces. ECG criteria suggesting epicardial surface will also be considered to define the epi or endo surface to be ablated.

Following ablation, a repeated programmed ventricular stimulation with S4 will be performed to evaluated reinducibility of the VT. Additional RF applications can be performed according to clinical criteria, and the procedure will be considered terminate when no VT is inducible or by clinical criteria. In the endo only group that endocardial scar could not be observed or following extensive endocardial ablation the clinical VT still remain inducible, and the ECG criteria suggests epicardial VT will underwent epicardial mapping and ablation and this will be considered as a Cross-over.

Outcomes

Primary Outcome:

Safety: The investigators will evaluate the rate of complications related to irrigated tip catheter use on epicardial surface. It is expected that the combined epicardial and endocardial ablation group do not present an increase in the rate of catheter-related complications.

Efficacy: The investigators will evaluate if the procedure was succeeded. The investigators consider success as follows: (1) Complete Success: prevention of induction of any VT following ablation; (2) Partial Success: prevention of induction of the clinical VT, remaining the induction of at least one non-clinical faster VT; (3) Failure: Remaining the induction of the clinical or initially induced VT.

Secondary Outcome:

Safety: The investigators will evaluate the rate of complications related to the epicardial access. It is expected a rate of hemopericardium of no more than 20%, with less than 5% rate of major complications as procedure related death, cardiac surgery due to cardiac perforation or blood cell transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic and non-ischemic cardiomyopathy and recurrent sustained monomorphic VT requiring cardioversion or antiarrhythmic drug administration with ≥4 episodes in the previous 6 months despite an ICD or antiarrhythmic drug therapy.
* Patients without ICD were eligible after 2 episodes of sustained VT.

Exclusion Criteria:

* Creatinine level >2.5mg/dL
* LV ejection fraction <10%
* NYHA Class IV
* Mobile thrombus on LV
* Absence of vascular access to the LV
* Life-expectancy of less than 12 months
* Previous open-chest cardiac surgical procedure
* Unstable angina; myocardial infarction in the last 2 months
* Severe aortic stenosis
* Severe mitral regurgitation secondary to leaflet or chordae rupture
* Pregnancy and age of less than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of epicardial ablation | Programed ventricular stimulation performed 5 minutes after complete ablation
  We will evaluate if the procedure was succeeded according to reinducibility of ventricular tachycardia. We consider success as follows: (1) Complete Success: prevention of induction of any VT following ablation; (2) Partial Success: prevention of induction of the clinical VT, remaining the induction of at least one non-clinical faster VT; (3) Failure: Remaining the induction of the clinical or initially induced VT.

SECONDARY OUTCOMES:
Safety of epicardial access | 24 hours after the procedure
  We will evaluate the rate of complications related to the epicardial access.
Safety of epicardial ablation using irrigated contact sensor catheter | At the end of the procedure
  We will evaluate the rate of complications related to irrigated tip catheter use on epicardial surface.

CONTACTS AND LOCATIONS:
Overall Officials: Maurício Scanavacca, MD, PhD, Principal Investigator — Instituto do coração - HC/FMUSP
Locations (1):
- Arrhythmia Clinical Unit - Instituto do Coração - HCFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pisani CF, Romero J, Lara S, Hardy C, Chokr M, Sacilotto L, Wu TC, Darrieux F, Hachul D, Kalil-Filho R, Di Biase L, Scanavacca M. Efficacy and safety of combined endocardial/epicardial catheter ablation for ventricular tachycardia in Chagas disease: A randomized controlled study. Heart Rhythm. 2020 Sep;17(9):1510-1518. doi: 10.1016/j.hrthm.2020.02.009. Epub 2020 Feb 20. PMID 32087356